CLINICAL TRIAL: NCT07080463
Title: Application of VascuLens 2.0, A Mixed Reality System for Surgical Guidance During DIEP Flap Harvest: A Randomized Controlled Trial
Acronym: VascuLens RCT
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kathryn Isaac, Assistant Professor and Surgeon, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H24-02372
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Vasculens

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- not using vasculens (No Intervention)
- using vasculens (Experimental)
  Interventions: Procedure: vasculens and cta

INTERVENTIONS:
Procedure: vasculens and cta — using vasculens and cta for one group and cta for the second group (control)
  Arms: using vasculens

SUMMARY:
This study incorporates the use of the VascuLens system, which relies on a mixed reality headset and software system, during the pre-operative stage of DIEP flap surgery. VascuLens utilizes augmented reality (AR) technology to project vasculature images obtained from computed tomography angiography (CTA) onto the patient's body. These projections are then traced onto the patient, and the accuracy of the key vascular anatomical landmarks in the projected images is compared to the accuracy of the conventional surgical markings of the same anatomical landmarks against the actual location of the dissected blood vessels. Higher accuracy may lead to improved patient care, reduced operative time and reduced risk of complications.

DETAILED DESCRIPTION:
Background and Rationale:

Breast reconstruction surgery is a surgical procedure that can be done after a breast removal surgery ("mastectomy"). One of the more common surgical methods for reconstruction involves taking a section of tissue from the abdomen that includes skin, fat, and blood vessels and relocating it to form the breast mound. This specific surgical method uses a section of the abdomen called the Deep Inferior Epigastric Artery Perforator (DIEP) flap. In order to accurately identify the necessary blood vessels for this surgery, surgeons generally take CTA (computed tomography angiography, a type of medical imaging to visualize a patient's blood vessels and tissues) of the abdomen before surgery to map out and visualize the positions of all the blood vessels during surgery.

The VascuLens is a mixed reality system that projects anatomical information onto a patient. In this study, the Vasculens system will project anatomical information, derived from the computed tomography angiography (CTA) images taken before surgery, onto a patient's body just prior to surgery.

In turn, the relevant projected vascular anatomy will be drawn onto the patient with a permanent marker. This will allow surgeons to see where important blood vessels are throughout the entire surgery rather than visualizing them in their minds. Great care, and a significant amount of time in the 8-hour DIEP flap reconstruction surgery, is often dedicated to separating the perforator arteries of the deep inferior epigastric artery and vein surrounding the rectus abdominis muscle. The authors of this study have developed the Vasculens system because they believe it will reduce the time to dissect the perforator arteries. Our pilot work confirmed the feasibility of use of the Vasculens system to accurately project patient-specific segmented anatomy for a DIEP free flap surgery.

Purpose:

The purpose of this study is to determine operative times with the use of the VascuLens system in comparison to the standard use of CTA in breast reconstruction with a DIEP flap. The standard of care for DIEP flap reconstruction is to obtain a preoperative CTA of the abdomen. These CTA images are reviewed pre-operatively and anatomic information is marked onto the patient using a ruler and marker for surgical planning. These are the standard surgical markings. In this study intervention, by using VascuLens, the CTA images and anatomic information will be projected onto the patient and traced onto the patient using a marker for surgical planning. The difference in standard of care is the additional visualization of the anatomic information being projected with use of VascuLens.

Objectives:

Primary Aims -To determine if use of the VascuLens system, a software using a mixed reality headset, reduces operative time for DIEP flap reconstruction surgery.

Secondary Aims

* To determine if use of the VascuLens system reduces surgical complications following DIEP flap reconstruction surgery.
* To determine if use of the VascuLens system reduces operative time variability for DIEP flap reconstruction surgery

Hypothesis:

Use of the VascuLens system reduces operative time and complications.

Study Design:

This is a randomized controlled trial with two parallel groups.The group allocation ratio for each study arm is 1:1.

* Group 1 (Control): Standard of care with DIEP flap harvest informed by CTA imaging only.
* Group 2 (Intervention): Standard of care with DIEP flap harvest informed by CTA imaging + VascuLens system.

This study occurs during all clinical visits which are part of standard of care, so no additional visits are required. The procedure occurs during the pre-operative and operative procedure and takes approximately 10 to 15 minutes during each stage.

Data Collection and Measures

There are TWO components to this study:

1. Operative times
2. Chart review of surgical complications

1. Operative Times

Operative times of the DIEP flap harvest will be collected by a research team member. Time points collected will be:

* Start of procedure, as determined by initial skin incision
* Identification of first perforator.
* perforator dissection.
* pedicle dissection.
* Flap harvest completion.
* The time from skin incision to completion of flap harvest will be the total procedure time.

  2. Surgical Complications
* Will be measured by abdominal bulge/hernia [Yes or No] recorded at 6 months, need to return to operating room and indication [yes or no, indications include arterial compromise, venous compromise, pedicle distortion, hematoma, thrombus], flap loss [Yes or No, partial or full], abdominal dehiscence, perforator injury, all recorded at 1 month post-operation. The chart review of this data will be collected by a research team member through participants' chart and EMR.

Additional data variables collected for assessment of potential confounders includes:

* Patient characteristics (BMI, age, surgical indication (immediate reconstruction, delayed reconstruction, delayed immediate reconstruction)
* Flap characteristics (number of perforators in harvested flap, flap volume)

Data Analysis:

Descriptive Statistics will be employed to present baseline patient characteristics (age, BMI, comorbidities) for both groups using means (SD) for continuous variables and frequencies (percentages) for categorical variables. Surgical Time will also be presented with descriptive statistics (mean, standard deviation, median, interquartile range) for surgical time in both groups.

Comparison of the primary outcome of surgical times will be completed by two-sample t-test (if the data is normally distributed) or Mann-Whitney U test (if data is non-normally distributed) for comparing the surgical times between the two groups. Normality of surgical times will be completed using the Shapiro-Wilk test. If the assumption of normality is violated, non-parametric tests will be selected. The effect size (Cohen's d) will be reported to quantify the magnitude of the difference in surgical times between the two groups.

Subgroup Analyses will be conducted based on factors including surgeon performing procedure, complexity of the surgery (number of perforators), and patient characteristics (BMI and flap volume).

For comparison of secondary outcomes, including complication rates, chi-squared test will be employed for categorical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 19 years old
* Patients must be undergoing a DIEP flap surgery after mastectomy for breast cancer or risk reduction
* Patient is already scheduled for a pre-operative CTA as part of routine standard of care.

Note: Non-English speaking participants will be given the option to have a translator.

Exclusion Criteria:

* Patients who have had a prior DIEP flap, as they may not have standard vascular anatomy and the previous surgery may have resulted in scarring and fibrosis that would potentially interfere with the accuracy of the projected anatomical information.
* Patients who have not had a pre-operative CTA because no imaging-based surgical guidance can be provided
* Patients who are pregnant at the time of surgery
* Patients who had a pre-operative CTA done before they were considered for this trial

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Operative times | surgery time

SECONDARY OUTCOMES:
Chart review of surgical complications | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UBC Breast Reconstruction Research Lab, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No